CLINICAL TRIAL: NCT01110083
Title: A Phase I Open-label, Non-randomized, Dose-escalation First-in-man Trial to Investigate the c-Met Kinase Inhibitor EMD 1204831 in Subjects With Advanced Solid Tumors
Brief Title: First-in-Man, Dose-escalation Trial of c-Met Kinase Inhibitor EMD 1204831 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Please see "Purpose" statement below.
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR200096-001
Record Dates: First submitted 2010-04-19; First posted 2010-04-26 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Solid Tumors
Keywords: Phase 1; advanced solid tumors; refractory to standard therapy; Patients with solid tumors, either refractory to standard therapy or for which no effective standard therapy is available
MeSH Terms: interventions — 4-(2-(2-(3-(3-(1-methyl-1H-pyrazol-4-yl)-6-oxo-1,6-dihydropyridazin-1-ylmethyl)phenyl)pyrimidin-5-yloxy)ethyl)morpholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: EMD 1204831

INTERVENTIONS:
Drug: EMD 1204831 — Subjects will receive EMD 1204831 twice a day for 21 days during each treatment cycle

SUMMARY:
EMD Serono has closed enrollment into this trial prior to determination of maximum tolerated dose (MTD). EMD Serono has decided not to pursue the development of EMD 1204831 in patients with advanced solid tumors for reasons other than safety.

DETAILED DESCRIPTION:
This is a an open-label, dose-escalation, first-in-man (FIM) study designed to explore the safety, tolerability, pharmacokinetics, and clinical activity of an investigational drug, EMD 1204831, in patients with advanced solid tumors who have not responded to previous therapies or for whom no other therapies are available. Subjects will receive EMD 1204831 twice a day (BID) during each 21-day cycle until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria

1. Histologically or cytologically confirmed solid tumor, either refractory standard therapy or for which no effective standard therapy is available
2. Measurable or evaluable disease, as defined by RECIST 1.0
3. Men or women aged ≥ 18 years
4. ECOG performance status of 0 to 2
5. Adequate hematological function: Hemoglobin ≥ 9.0 g/dL; Neutrophils > 1.5 x 109/L; Platelets ≥ 100 x 109/L
6. Adequate liver function: Total bilirubin ≤ 1.5 x ULN; AST/ ALT ≤ 2.5 x ULN
7. For subjects with liver metastases: Total bilirubin ≤ 1.5 x ULN; AST/ALT ≤ 5 ULN
8. Adequate renal function: Serum creatinine < 1.5 x ULN, and/or Calculated creatinine clearance > 60 mL/min
9. Resolution of all acute chemotherapy, radiotherapy or surgery-related AEs to Grade ≤1, except for alopecia
10. Recovery from any surgical intervention
11. Subjects enrolling after the MTD has been determined must present specific c-Met alterations (overexpression, amplification, mutation)

Exclusion Criteria:

Main Exclusion Criteria

1. Received chemotherapy, immunotherapy, hormonal therapy (except subjects with prostate cancer), biologic therapy, or any other investigational agent or anticancer therapy within 28 days (or five half-lives for non-cytotoxics, whichever is shorter), of Day 1 of trial treatment (six weeks for nitrosureas or mitomycin C)
2. Received extensive prior radiotherapy on more than 30% of bone marrow
3. Symptomatic primary tumors or metastasis of brain and/or central nervous system, uncontrolled with antiepileptics and requiring high doses of steroids
4. Medical history of liver fibrosis/ cirrhosis
5. Medical history of surgery within six weeks prior to enrollment
6. Neuropathy Grade ≥ 2
7. Requires concurrent treatment with a non-permitted drug
8. Absence or abnormal pupillary reflex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of EMD 1204831 in subjects with advanced solid tumors | After first cycle of treatment

SECONDARY OUTCOMES:
Number and frequency of adverse events, and changes from baseline in laboratory values, vital signs and ECGs will be used to assess safety and tolerability of EMD1204831. | Scheduled visits throuhout each 21 day cycle of treatment. Subjects may continue to receive cycles of EMD 1204831 until disease progression or unacceptable toxicity.
Anti-tumor activity and best overall response will be assessed according to RECIST 1.0 after every two cycles of EMD 1204831. Frequency of subjects with different levels of overall response (CR, PR, SD or PD) and best Overall Response will be presented. | Scheduled visits throuhout each 21 day cycle of treatment. Subjects may continue to receive cycles of EMD 1204831 until disease progression or unacceptable toxicity.
PK parameters will be assessed to characterize the pharmacokinetic (PK) profile of EMD 1204831 and summarized by dose level and cycle. | Scheduled visits throuhout each 21 day cycle of treatment. Subjects may continue to receive cycles of EMD 1204831 until disease progression or unacceptable toxicity.
Values and changes over time in pharmacodynamic (Pd) markers in tissue and molecular markers in blood will be assessed | Scheduled visits throuhout each 21 day cycle of treatment. Subjects may continue to receive cycles of EMD 1204831 until disease progression or unacceptable toxicity.
Exploratory analyses of genes that may be involved in the absorption, distribution, metabolism, and elimination (ADME) of EMD 1204831 will be performed. | Scheduled visits throuhout each 21 day cycle of treatment. Subjects may continue to receive cycles of EMD 1204831 until disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Klevasath, MD, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States